CLINICAL TRIAL: NCT02490722
Title: The Effect of Interdisciplinary Group Based Patient Education on Functions in Patients With Non-specific and/or Degenerative Low Back Pain
Brief Title: Effect of Patient Education on Functions in Patients With Non-specific and/or Degenerative Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-15006949
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2017-07

CONDITIONS: Low Back Pain
Keywords: Patient education; Empowerment
MeSH Terms: conditions — Low Back Pain; Empowerment | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Four times two hours interdisciplinary patient education and usual care
  Interventions: Other: Patient education
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Patient education — Four times two hours group based patient education
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate effects of interdisciplinary group based patient education in patients with low back pain.

The patients will be recruited to four group based patient education lessons during a two months period. The study is a randomized controlled trial and the patients will be randomized to standard treatment or standard treatment and patient education. The patient education will be led by physiotherapists, nurses and physicians. The outcomes are functions, pain, quality of life, self-efficacy, and depression. The data are reported in questionnaires.

DETAILED DESCRIPTION:
Design: Randomized controlled trial; intervention study. Patients: Patients with low back pain; referred to Nordsjaellands Hospital, Denmark. Inclusion criteria: adults, low back pain minimum scored 4 on numeric rating scale, able to conduct exercise training. Exclusion criteria: unable to understand Danish, psychiatric disorder, dementia, approaching operation, current or approaching settlement regarding working ability or compensation as a result of low back pain. Intervention: Randomization to usual care or usual care and four times two hours group based patient education with an interdisciplinary focus on self-management of low back pain. The patient education will be delivered by physiotherapists, nurses and physicians. Outcome: functions, pain, quality of life, self-efficacy, and depression. The data are reported in questionnaires. Sample size: 74 participants.

ELIGIBILITY:
Inclusion Criteria:

* adults
* low back pain minimum scored 4 on numeric rating scale
* able to conduct exercise training

Exclusion Criteria:

* unable to understand Danish
* psychiatric disorder
* dementia
* approaching operation
* current or approaching settlement regarding working ability or compensation as a result of low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change of functions | Patients will be followed for a period of two months with four patients education sessions. Follow-up will be tested 12 weeks after the last education session.
  Questionnaire

SECONDARY OUTCOMES:
Change of pain | Patients will be followed for a period of two months with four patients education sessions. Follow-up will be tested 12 weeks after the last education session.
  Questionnaire
Change of self-efficacy | Patients will be followed for a period of two months with four patients education sessions. Follow-up will be tested 12 weeks after the last education session.
  Questionnaire
Change of quality of life | Patients will be followed for a period of two months with four patients education sessions. Follow-up will be tested 12 weeks after the last education session.
  Questionnaire
Change of depression | Patients will be followed for a period of two months with four patients education sessions. Follow-up will be tested 12 weeks after the last education session.
  Questionnaire
Change of physical function | Patients will be followed for a period of two months with four patients education sessions. Follow-up will be tested 12 weeks after the last education session.
  Performance test

CONTACTS AND LOCATIONS:
Overall Officials: Stig Molsted, PhD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heymans MW, van Tulder MW, Esmail R, Bombardier C, Koes BW. Back schools for non-specific low-back pain. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD000261. doi: 10.1002/14651858.CD000261.pub2. PMID 15494995
- [Background] Dufour N, Thamsborg G, Oefeldt A, Lundsgaard C, Stender S. Treatment of chronic low back pain: a randomized, clinical trial comparing group-based multidisciplinary biopsychosocial rehabilitation and intensive individual therapist-assisted back muscle strengthening exercises. Spine (Phila Pa 1976). 2010 Mar 1;35(5):469-76. doi: 10.1097/BRS.0b013e3181b8db2e. PMID 20147878
- [Background] Morone G, Paolucci T, Alcuri MR, Vulpiani MC, Matano A, Bureca I, Paolucci S, Saraceni VM. Quality of life improved by multidisciplinary back school program in patients with chronic non-specific low back pain: a single blind randomized controlled trial. Eur J Phys Rehabil Med. 2011 Dec;47(4):533-41. Epub 2011 Apr 20. PMID 21508915